CLINICAL TRIAL: NCT01062295
Title: Efficacy and Safety of the Device Siesta-SystemTM for Inducing Objective Sleep and re Rest.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Joaquin Duran-Cantolla, Osakidetza/Basque Health Service
Model: Crossover | Purpose: Supportive Care
Other Study IDs: conductores
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2009-10

CONDITIONS: Sleep
Keywords: passenger,; sleep,; rest,

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Siesta-System (Experimental): Use of Siesta-System
  Interventions: Device: Siesta-System
- Standard headrest (Active Comparator): Use of standard headrest
  Interventions: Device: Standard headrest

INTERVENTIONS:
Device: Siesta-System
  Arms: Siesta-System
Device: Standard headrest
  Arms: Standard headrest

SUMMARY:
NTRODUCTION: The investigators have developed a new device to help passengers of vehicles to rest, sleep, and to avoid cervical injuries due to sleepiness postures while travelling. The device is attached to the headrest and is based in a new concept called "dynamic vertical holding of the head and neck". It could also provide some help in avoiding accidents by allowing a sleeping time for a secondary driver while the main one is driving. Several studies have shown that up to 30% of car crashes are related to sleepiness.

AIM: To estimate the efficacy and safety of a new device in "patent pending" phase to facilitate the sleep and rest in the passenger.

METODOLOGY: DESIGN: Prospective, cross-over and open clinical assay, comparing the results of 40 different passengers during a journey after using both systems, that is the new device and the standard headrest.

MEASUREMENTS: A) Standard polysomnography for 3 and a half hours during the night; B) Anthropometric and clinical variables; C) Sleepiness scale and Epworth sleepiness; D) Questionnaires of sleep, health and quality of life. E) Evaluation of the neck posture in recorded images.

ANALYSIS: To compare the results of questionnaires of sleep quality, comfort and safety as well as the images recorded and polysomnographic variables of objective sleep variables obtained by the device Siesta-SystemTM and the conventional headrest.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 30 and 80 years

Exclusion Criteria:

* People with back pain or hip area on trips of 5 hours. Acute passenger. Serious chronic illness. Depressions. Medicated people with sleep inducing drugs or stimulants. People with insomnia relevant and apnea-hypopnea syndrome during sleep (SAHS) will be excluded by validated sleep test. People who have drunk in the last 6 hours coffee, other drinks, exciting, or an amount of alcohol over a glass of wine and those who stayed more than 30 minutes las12 hours before the test. People who declare themselves unable to relax in a vehicle while riding as co-pilots. Morbid obesity (BMI> 40 kg/m2) and any musculoskeletal disorder defined as a disease that can trouble the rest and sleep onset in a car. Latex allergy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2009-05 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Durán-Cantolla, MD, PhD, Principal Investigator — Osakidetza/ Basque Health System
Locations (1):
- Txagorritxu Hospital, Vitoria-Gasteiz, Alava, Spain

REFERENCES:
- [Derived] Lopez-Valdes FJ, Fernandez-Bolanos Martin M, Alvarez Ruiz-Larrinaga A, Segui-Gomez M. Reduction in the exposure to being out-of-position among car occupants who used a sleeping device. Inj Prev. 2012 Jun;18(3):165-9. doi: 10.1136/injuryprev-2011-040031. Epub 2011 Sep 8. PMID 21903969